CLINICAL TRIAL: NCT03791008
Title: Personalized Breast Cancer Screening: Assessment of Its Feasibility and Acceptability in the National Health System
Brief Title: Assessment of Feasibility and Acceptability of Personalized Breast Cancer Screening
Acronym: DECIDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recerca Biomèdica de Lleida (Other)
Collaborators: Institut Català de la Salut (Other); Catalan Health Service (Unknown)
Responsible Party: Principal Investigator, Montserrat Rue, Professor, Institut de Recerca Biomèdica de Lleida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PI17/00834
Record Dates: First submitted 2018-11-16; First posted 2019-01-02 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer
Keywords: Personalized; Early detection; Screening; Feasibility; Acceptability
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Risk based screening — Breast cancer risk measurement, screening recommendations and shared decision making

SUMMARY:
The overall objective is to assess the acceptability and feasibility of offering personalized breast cancer (BC) screening.

The specific objectives are: 1) To design an information system; 2) To evaluate the barriers and facilitators of the coordination of health care services and the screening program; 3) To develop a proof of concept of personalized screening; and 4) To evaluate cost-effectiveness.

Methodology:

1. Prototype information system with basal and longitudinal variables relevant to a personalized screening system;
2. Qualitative study with focus groups and survey. The attitude and acceptability on a sample of 210 health professionals will be assessed;
3. Prospective observational study, for proof of concept. Participants will be professionals working in Primary Care, Population Breast Screening Program, or Hospital Breast Unit. It will include 385 women, aged 40-50 from the city of Lleida. Various indicators of acceptability and feasibility will be assessed in women and health professionals;
4. Probabilistic analytical models will be used to evaluate cost-effectiveness.

The present protocol addresses the specific objective number 3, the proof of concept of personalised screening.

Expected results: The investigators expect to provide valuable and necessary information for the design of personalized screening.

ELIGIBILITY:
Inclusion Criteria:

* Not having had a mammogram in the last 12 months or with a mammogram in this period available to evaluate breast density.
* Sign the informed consent.

Exclusion Criteria:

* Previous diagnosis of breast cancer.
* Breast study in process.
* Fulfill clinical criteria defined by the Medical Oncology Spanish Society (SEOM to refer to the genetic counseling unit in cancer.
* Do not understand or speak Catalan or Spanish.
* Cognitive disability for mental or mental illness.
* Physical disability that prevents a mammogram.

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 387 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Attitude towards personalised breast cancer screening (by participant women) | 2-4 weeks after being informed of the individual breast cancer risk
  Attitude scale with three items, one about the frequency of screening exams (ranges from 1 to 5). The other two items ask if participants are satisfied of being invited more/less frequently, in case that they have a higher/lower risk of breast cancer than the average women. They also range from 1 to 5. Total scores can range from 3 to 15. Higher scores indicate more positive attitudes. A positive attitude is defined as a total score greater or equal to 12. Adapted from Hersch et al. (2015)
Intention to participate in personalised breast cancer screening | 2-4 weeks after being informed of the individual breast cancer risk
  Categorical variable with five categories: definitely will, likely to, unsure, not likely to, definitely will not. The absolute and relative frequencies of the five categories will be obtained. In addition, the variable will be dichotomized as intending to participate (definitely or likely) or not. Adapted from Hersch et al. (2015)
Satisfaction with personalised screening | At 1 year of the study start
  Satisfaction Likert scale with one item that ranges from 1 to 5: not at all satisfied (1), extremely satisfied (5). Following the Sekhon et al. review (2017)

SECONDARY OUTCOMES:
Screening attitudes scale | 2-4 weeks after being informed of the individual breast cancer risk
  General attitudes scale towards screening mammography. It will be measured using five items adapted from Hersch et al. (2015). Each item ranges from 1 to 5. Total scores can range from 5 to 25. A positive attitude is defined as a total score greater or equal to 20. Higher scores indicate more positive attitudes. Adapted from Hersch et al. (2015)
Attitude towards the measure of breast cancer risk | 2-4 weeks after being informed of the individual breast cancer risk
  One categorical variable with four categories. It asks if the measure of breast cancer risk will do more harm than good, more good than harm, it depends, do not know. The absolute and relative frequencies of the four categories will be obtained. Following the Sekhon et al. review (2017)
Emotional impact of the measure of breast cancer risk | 2-4 weeks after being informed of the individual breast cancer risk
  Three categorical variables with five categories, ranging from strongly disagree (1) to strongly agree (5). First variable: The information about the individual risk of breast cancer provides calmness. Second variable: Receiving information about risks produces anxiety. Third variable: The information about the individual risk of breast cancer makes me worry. The scores of the three items will not be added as a scale, they will be reported separately. Adapted from Hersch et al. (2015)
Preference with regard to the current screening, biennial between 50 and 69 years | 2-4 weeks after being informed of the individual breast cancer risk
  Categorical variable with three categories. It asks what type of screening the participants would choose (personalized risk-based or "one-size-fits-all")
Knowledge of the benefits and harms of breast cancer screening | 2-4 weeks after being informed of the individual breast cancer risk
  Eleven conceptual knowledge questions (Yes/No) and four numerical knowledge questions with categories on the effect of screening. A total of 22 marks could be obtained, 11 coming from the questions on conceptual knowledge and 11 coming from the questions on numerical knowledge that measured absolute and relative values of the screening outcomes. The threshold to define adequate knowledge is to score at least 50% of the available marks, including at least one numerical mark, on all the three screening outcome subscales that refer to mortality reduction, overdiagnosis, and false positives. Adapted from Hersch et al. (2015)
Decisional conflict | 2-4 weeks after being informed of the individual breast cancer risk
  O'Connor Decisional Conflict Scale, 10-item low literacy version, on a scale from 0 (no decisional conflict) to 100 (extreme decisional conflict). Scores less than 25 are associated with implementing decisions; score exceeding 37.5 are associated with decision delay or feeling unsure about implementation.
Confidence in the decision | 2-4 weeks after being informed of the individual breast cancer risk
  Three Likert scale statements rated from 1 (not at all confident) to 5 (very confident). A total score is obtained summing the scores of the three items and dividing by three.
  Adapted from the O'Connor Decision Self-Efficacy Scale
Anxiety about screening participation | 2-4 weeks after being informed of the individual breast cancer risk
  Six-item short form of the Spielberger State Trait Anxiety Inventory (STAI) on a scale from 20 to 80, with higher scores indicating greater levels of anxiety. To calculate the total STAI score, reverse scoring of the positive items (calm, relaxed, content), sum all six scores and multiply total score by 20/6.
Perceived significance of the benefits and the adverse effects of screening | 2-4 weeks after being informed of the individual breast cancer risk
  Women will be asked how important it is for them to consider the chances of (1) avoiding breast cancer death, (2) being diagnosed and treated for a cancer that is not harmful, and (3) having a false positive. The four response options range from very important (1) to not at all important (4). The scores of the three items will not be added as a scale, they will be reported separately. According to Hersch et al. (2015)
Self-efficacy | 2-4 weeks after being informed of the individual breast cancer risk
  Four items ranging from strongly disagree (1) to strongly agree (5). Total scores can range from 4 to 20. Higher scores indicate higher self-efficacy. Following the Sekhon et al. review (2017)
Experience assessment | 2-4 weeks after being informed of the individual breast cancer risk
  It will be measured using five items. Each item ranges from 1 to 5. Total scores can range from 5 to 25. A positive assessment is defined as a total score greater or equal to 20. Higher scores indicate more positive experience assessment. Following the Sekhon et al. review (2017)
Confidence in personalised screening | 2-4 weeks after being informed of the individual breast cancer risk
  Confidence Likert scale with one item ranging from very low confidence (1) to very high confidence (5) . Following the Sekhon et al. review (2017)
Understanding of the individual risk and the screening recommendations | 2-4 weeks after being informed of the individual breast cancer risk
  Two categorical variables with five categories each, ranging from strongly disagree (1) to strongly agree (5). First variable: I understood the information I received about my risk of breast cancer in relation to women of my age. Second variable: I have understood the recommendations given to me about the screening of breast cancer in the coming years, based on my risk of breast cancer. The scores of the two items will not be added as a scale, they will be reported separately. Following the Sekhon et al. review (2017)
Time spent on risk communication | At the time of communicating risk, 2-4 weeks after the baseline visit
  Continuous variable, number of minutes. Recorded by the participant doctors
Proportion of women who accept to participate in the study | Through study completion, an average of 1.75 years
  Number of women that accept to participate divided by number of women contacted
Proportion of participating women who complete the different phases of the study | Through study completion, an average of 1.75 years
  Number of women that complete the different phases divided by number of participating women

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recerca Biomèdica de Lleida, Lleida, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hersch J, Barratt A, Jansen J, Irwig L, McGeechan K, Jacklyn G, Thornton H, Dhillon H, Houssami N, McCaffery K. Use of a decision aid including information on overdetection to support informed choice about breast cancer screening: a randomised controlled trial. Lancet. 2015 Apr 25;385(9978):1642-52. doi: 10.1016/S0140-6736(15)60123-4. Epub 2015 Feb 18. PMID 25701273
- [Background] Sekhon M, Cartwright M, Francis JJ. Acceptability of healthcare interventions: an overview of reviews and development of a theoretical framework. BMC Health Serv Res. 2017 Jan 26;17(1):88. doi: 10.1186/s12913-017-2031-8. PMID 28126032
- [Derived] Pons-Rodriguez A, Forne Izquierdo C, Vilaplana-Mayoral J, Cruz-Esteve I, Sanchez-Lopez I, Rene-Rene M, Cazorla C, Hernandez-Andreu M, Galindo-Ortego G, Llorens Gabande M, Laza-Vasquez C, Balaguer-Llaquet P, Martinez-Alonso M, Rue M; DECIDO Group. Feasibility and acceptability of personalised breast cancer screening (DECIDO study): protocol of a single-arm proof-of-concept trial. BMJ Open. 2020 Dec 23;10(12):e044597. doi: 10.1136/bmjopen-2020-044597. PMID 33361170